CLINICAL TRIAL: NCT02041780
Title: Non Invasive Assessment of Liver Fibrosis in Children: Evaluation of Diagnostic Performances of ShearWave Elastography (SWE) and Fibrotest®/ Fibromax® by Comparison With Fibrosis Score on Liver Biopsy
Brief Title: Non Invasive Assessment of Liver Fibrosis in Children: Comparison of ShearWave Elastography, Fibrotest and Liver Biopsy
Acronym: SHEARWAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120128
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Liver Fibrosis; Children
Keywords: Diagnostic; Liver fibrosis; Ishak score; Fibrotest; ShearWave elastography; Liver biopsies
MeSH Terms: conditions — Liver Cirrhosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shearwave electrography (Experimental): Two experimental interventions will be realized in each patient in this population : Shearwave electrography (new diagnostic test of fibrosis) and Fibrotest .
  Moreover, liver biopsies, the gold standard for the fibrosis diagnosis is also realized in each patient within usual cares.
  Interventions: Procedure: Shearwave electrography

INTERVENTIONS:
Procedure: Shearwave electrography

SUMMARY:
The purpose of this study is to determine if SWE and Fibrotest®/ Fibromax®, alone or associated, are effective methods to assess liver fibrosis in children.

DETAILED DESCRIPTION:
Liver biopsy will be the gold standard to assess fibrosis using Ishak score and morphometric evaluation of fibrosis. All children included will have a measure of liver stiffness using SWE with 5 measures performed in the area where the biopsy is performed and 5 measures in an other place in the liver. Fibrotest®/ Fibromax® will be performed on blood sample. All exams will be done within 1 month. diagnostic performance of SWE and Fibrotest®/ Fibromax® will be assessed respectively. algorithm using the results of both technics will be tested in order to test diagnostic performance and to obtain better performances.

ELIGIBILITY:
Inclusion Criteria:

* age < 18 years;
* indication to liver biopsy;
* informed consent of both parents and child if applicable;
* social insurance

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
liver fibrosis evaluated by the ISHAK score and morphometric evaluation | up to 1 month
  Histology is the gold standard to evaluate liver fibrosis

SECONDARY OUTCOMES:
liver fibrosis evaluation : stiffness using SHEARWAVE elastography | up 1 month
Liver fibrosis evaluation using Fibrotest (Fibromax) | up 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie FRANCHI-ABELA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France